CLINICAL TRIAL: NCT07222917
Title: A Phase IIb, Randomised, Multicentre, Double-Blind Study to Evaluate the Effect of Baxdrostat in Combination With Dapagliflozin Compared With Baxdrostat on Albuminuria in Participants With Chronic Kidney Disease and High Blood Pressure.
Brief Title: A Phase IIb Study to Evaluate the Effect of Dapagliflozin in Combination With Baxdrostat Compared With Baxdrostat on Albuminuria in Participants With Chronic Kidney Disease and High Blood Pressure.
Acronym: BaxDuo-Baltic
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6972C00006
Record Dates: First submitted 2025-10-17; First posted 2025-10-30 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease and Hypertension
Keywords: Chronic kidney disease; Hypertension; Blood pressure; Baxdrostat; Dapagliflozin
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Interventional, multicentre, randomised, double-blind, parallel group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The IRT/RTSM will provide to the Investigator(s) or pharmacist(s) the kit identification number to be allocated to the participant at the dispensing visit.
  The following personnel will be unblinded:
  * Personnel carrying out the packaging and labelling of study intervention treatment
  * Personnel generating the randomisation list
  Participants, site personnel, and AstraZeneca will be blinded to study intervention. AstraZeneca retains the right to break the code for SAEs that are unexpected and are suspected to be causally related to study intervention and that potentially require expedited reporting to regulatory authorities. Randomisation codes will not be broken for the planned analyses of data until all decisions on the evaluability of the data from each individual participant have been made and documented.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Baxdrostat/dapagliflozin (Experimental): Participants randomised to the baxdrostat/dapagliflozin arm will receive one dose of baxdrostat and one standard dose of dapagliflozin daily.
  Interventions: Drug: Baxdrostat/dapagliflozin
- Baxdrostat /placebo (Placebo Comparator): Patients will receive one dose of baxdrostat comparator in combination with placebo matching dapagliflozin daily
  Interventions: Drug: Baxdrostat/Placebo

INTERVENTIONS:
Drug: Baxdrostat/dapagliflozin — baxdrostat tablet
  dapagliflozin tablet
  Arms: Baxdrostat/dapagliflozin
Drug: Baxdrostat/Placebo — baxdrostat tablet
  placebo tablet
  Arms: Baxdrostat /placebo

SUMMARY:
International, Multicenter and Double-Blind study. The purpose is to measure the effect of baxdrostat in combination with dapagliflozin compared with baxdrostat/placebo on albuminuria, as well as safety, in participants with chronic kidney disease and high blood pressure.

DETAILED DESCRIPTION:
This is a Phase IIb, randomised, multicentre, double-blind, parallel-group study aiming to determine the effect on albuminuria, as well as safety, of baxdrostat/dapagliflozin compared with baxdrostat/placebo, when given to participants with CKD and high blood pressure.

Study population will include participants ≥ 18 years old with CKD. Participants with or without a diagnosis of T2DM and with or without an SGLT2i treatment at screening are eligible for the study.

The study will include an optional pre-screening period, where participants will be assessed for at least one of the following parameters: eGFR, UACR, potassium, sodium, and BP. Participants who are being treated with SGLT2i at the time of the screening visit will complete a washout period After screening and initial confirmation of eligibility, participants will be randomised to receive either baxdrostat/dapagliflozin or baxdrostat/placebo. For randomisation there will be stratification and capping linked to T2DM status.

The primary objective is to assess the effect of baxdrostat/dapagliflozin compared with baxdrostat/matching placebo on albuminuria, which will be evaluated by change from baseline in UACR.

The end of the study is defined as the date of the last visit of the last participant in the study or last scheduled procedure shown in the SoA for the last participant in the study globally, whichever occurs last.

A participant is considered to have completed the study if they have completed all periods of the study including the last scheduled procedure shown in the SoA.

ELIGIBILITY:
Inclusion Criteria:

1. Participants of any sex and gender must be ≥ 18 years of age at the time of signing the informed consent.
2. Participants with eGFR ≥ 30 and < 90 mL/min/1.73 m2 at screening
3. Participants with UACR > 200 mg/g (22.6 mg/mmol) and < 5000 mg/g (565 mg/mmol) at screening
4. Participants with history of HTN and a SBP ≥ 130 mmHg at screening and ≥ 120 mmHg at the randomisation visit.
5. Stable and maximum daily tolerated dose of either an ACE inhibitor or an ARB (not both) for at least 4 weeks prior to the screening visit, if not medically contraindicated.
6. Participants with:

   1. Serum or plasma potassium ≥ 3.0 and ≤ 4.8 mmol/L if eGFR ≥ 45 mL/min/1.73 m2.
   2. Serum or plasma potassium ≥ 3.0 and ≤ 4.5 mmol/L if eGFR < 45 mL/min/1.73 m2.
7. Contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. Applicable to female participants.

Exclusion Criteria:

1. Systolic blood pressure > 180 mmHg, or diastolic blood pressure > 110 mmHg at screening.
2. Known hyperkalaemia, defined as potassium of ≥ 5.5 mmol/L within 3 months before screening
3. Serum sodium < 135 mmol/L at the Screening Visit (values obtained within 4 weeks prior to screening or at the Screening Visit).
4. Diabetes mellitus:

   1. T1DM at the screening visit
   2. Uncontrolled T2DM at screening: HbA1C > 10.5% (> 91 mmol/mol)
5. New York Heart Association functional HF class IV at screening
6. Any use of mineralocorticoid receptor antagonists (such as spironolactone, eplerenone, or finerenone), aldosterone synthase inhibitors, potassium-sparing diuretics (such as triamterene or amiloride), or potassium binders (such as sodium zirconium cyclosilicate, patiromer, or sodium polystyrene sulfonate) within 4 weeks prior to screening
7. Stroke, transient ischaemic cerebral attack, valve implantation or valve replacement, carotid surgery, or carotid angioplasty, acute coronary syndrome, or hospitalisation for worsening HF within previous 3 months prior to randomisation.
8. Known severe hepatic impairment, defined as Child-Pugh Class C, based on records that confirm documented medical history.
9. Documented history of adrenal insufficiency.
10. Any dialysis (including for acute kidney injury) within 3 months prior to the screening
11. Any acute kidney injury within 3 months prior to the screening visit.
12. Prohibited concomitant medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2027-05-24 (Estimated); Study Completion 2027-05-24 (Estimated)

PRIMARY OUTCOMES:
To determine whether baxdrostat/dapagliflozin is superior to baxdrostat/matching placebo at reducing albuminuria. | Up to 12 weeks
  Change from baseline in UACR

CONTACTS AND LOCATIONS:
Locations (59):
- United States (18):
  - Research Site, Surprise, Arizona
  - Research Site, Hollywood, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Champaign, Illinois
  - Research Site, Wichita, Kansas
  - Research Site, Eatontown, New Jersey
  - Research Site, Greenville, North Carolina
  - Research Site, Jacksonville, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Media, Pennsylvania
  - Research Site, East Providence, Rhode Island
  - Research Site, Arlington, Texas
  - Research Site, Pasadena, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Woodbridge, Virginia
- Argentina (4):
  - Research Site, Buenos Aires
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Mar del Plata
  - Research Site, San Nicolás
- Bulgaria (4):
  - Research Site, Pernik
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Yambol
- Canada (5):
  - Research Site, Courtice, Ontario
  - Research Site, Etobicoke, Ontario
  - Research Site, Stouffville, Ontario
  - Research Site, Waterloo, Ontario
  - Research Site, Montreal, Quebec
- South Korea (4):
  - Research Site, Anyang-si
  - Research Site, Cheonan-si
  - Research Site, Goyang-si
  - Research Site, Seoul
- Spain (3):
  - Research Site, Badalona
  - Research Site, Pamplona
  - Research Site, Valencia
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (5):
  - Research Site, Bangkoknoi
  - Research Site, Changwat Sara Buri
  - Research Site, Hat Yai
  - Research Site, Muang
  - Research Site, Ratchathewi
- Turkey (Türkiye) (5):
  - Research Site, Adana
  - Research Site, Adapazarı
  - Research Site, Kahramanmaraş
  - Research Site, Kayseri
  - Research Site, Kocaeli
- Ukraine (3):
  - Research Site, Kyiv
  - Research Site, Uzhhorod
  - Research Site, Vinnytsia
- United Kingdom (3):
  - Research Site, Dundee
  - Research Site, Liverpool
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/